CLINICAL TRIAL: NCT05748262
Title: Department of Infectious Diseases, Shanghai Key Laboratory of Infectious Diseases and Biosafety Emergency Response, National Medical Center for Infectious Diseases, Huashan Hospital, Fudan University, Shanghai, China;
Brief Title: Characteristics of SARS-CoV-2 Reinfection
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Jiming Zhang (Other)
Responsible Party: Sponsor-Investigator, Jiming Zhang, professor, Huashan Hospital
Organization: Huashan Hospital (Other)
Other Study IDs: 2022-721
Record Dates: First submitted 2023-02-12; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: Reinfection; risk factor; clinical severity
MeSH Terms: conditions — COVID-19; Reinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary infections during March-May 2022: Hospitalized COVID-19 patients infected with BA·2 during 1 March to 23 May 2022 from Huashan Hospital, Renji Hospital, and Shanghai Jing' an Central Hospital.
- Primary infections during December 2022-January 2023: Primary infections with BA.5-sublineages during 1 December 2022 to 14 January 2023, matched 1:1 by age and sex with reinfections during the same period.

SUMMARY:
As the COVID-19 pandemic continues and the number of individuals with previous infection rises, numbers of SARS-CoV-2 reinfection are increasing. The second Omicron wave in Shanghai, China caused by BA.5-sublineages led to a large fraction of reinfections among BA.2 primary infections. To better understand the SARS-CoV-2 reinfection rate and clinical severity of reinfections, the investigators conducted a multi-centre cohort study. The investigators hope to provide valuable clinical evidences for reinfections and offer guidance for future policy making.

DETAILED DESCRIPTION:
The investigators used data from Huashan Hospital, Renji Hospital, and Shanghai Jing' an Central Hospital to collect information on SARS-CoV-2 primary infections with BA.2 during 1 March to 23 May 2022, and followed up for participants' reinfections with BA.5-lineages during 1 December 2022 to 14 January 2023. After matched 1:1 by age and gender with the reinfection cohort, data of primary infections with BA.5-sublineages were also collected. Reinfection cases were defined as having positive COVID-19 PCR or antigen test, at least 90 days after participants' first positive testing. Basic information, vaccination status, time interval between two infections, and clinical manifestations were collected.

ELIGIBILITY:
Inclusion Criteria:

* All PCR- or RAT-confirmed SARS-CoV-2 reinfections were included in the study.

Exclusion Criteria:

* Patients who did not know if they were reinfected were excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A Primary SARS-CoV-2 infection was defined as having a positive PCR test result for the first time. A suspect SARS-CoV-2 reinfection (generally referred as reinfection in this paper) was defined as having a positive PCR of RAT sample over 90 days following primary infection.
Sampling Method: Non-Probability Sample
Enrollment: 1144 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-03-20 (Estimated); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
Characteristics of all enrolled SARS-CoV-2 patients during two periods. | 2022-12~2023-2
  Basic information, vaccination status, time interval between two infections, and clinical manifestations
Characteristics and multivariate analysis of risk factors for SARS-CoV-2 reinfection by gender, age, vaccination status, clinical severity and Ct values of primary infection. | 2022-12~2023-2
  Sex, age, vaccination status, clinical severity of primary infection, and Ct values during primary infection
Clinical characteristics of SARS-CoV-2 primary infection and reinfection among patients with reinfection in Shanghai | 2022-12~2023-2
  Fever, fatigue, sore throat, cough, anosmia and/or ageusia, muscle and/or joint pain, headache, chest congestion, diarrhea, runny nose, sleeping disorders, and pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Jiming Zhang, PhD, Study Director — Huashan Hospital
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (including data dictionaries) will be available. Individual participant data that underlie the results reported in this article will be shared after de-identification (text, tables, figures, and appendices). Study protocol will also be available. The time period for data sharing begins nine months and ends 36 months following article publication. Data is available with investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our university's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at https://yxky.fudan.edu.cn.
Supporting Information: Study Protocol, SAP
Time Frame: The time period for data sharing begins nine months and ends 36 months following article publication.
Access Criteria: Data is available with investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for individual participant data meta-analysis.
URL: http://yxky.fudan.edu.cn